CLINICAL TRIAL: NCT00605631
Title: The Prevention of Myocardial Enlargement and Dilatation Post Myocardial Infarction Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MENDMI
Record Dates: First submitted 2007-12-20; First posted 2008-01-31 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Post Myocardial Infarction
Keywords: Pacing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Device: Cardiac pacing using any Guidant/Boston Scientific Implantable ICD or CRT-D System and any Guidant/Boston Scientific Intracardiac Lead System
- 2 (Active Comparator)
  Interventions: Device: Cardiac pacing using any Guidant/Boston Scientific Implantable ICD or CRT-D System and any Guidant/Boston Scientific Intracardiac Lead System
- 3 (Other)
  Interventions: Device: Cardiac pacing using any Guidant/Boston Scientific Implantable ICD or CRT-D System and any Guidant/Boston Scientific Intracardiac Lead System

INTERVENTIONS:
Device: Cardiac pacing using any Guidant/Boston Scientific Implantable ICD or CRT-D System and any Guidant/Boston Scientific Intracardiac Lead System — No specific device model is required - any FDA-approved, market-released Guidant/Boston Scientific implantable ICD or CRT-D system and any FDA-approved, market-released Guidant/Boston Scientific intracardiac lead system may be implanted as part of MENDMI.

SUMMARY:
This study is designed to evaluate the effect of pacing on post-MI patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above, or of legal age to give informed consent specific to state and national law
* Willing and capable of providing informed consent, participating in all testing associated with this clinical investigation at an approved clinical investigational center and at the intervals defined by this protocol
* Patient has had a clinically documented anterior myocardial infarction which occurred within the last 14 days
* Measured peak CK > 2000 mU/mL within 72 hours of MI.
* QRS duration < 120 ms measured by 12-lead ECG at any time after most recent MI

Exclusion Criteria:

* Patient has atrial tachyarrhythmia that is permanent (i.e., does not terminate spontaneously and cannot be terminated with medical intervention) or persistent (i.e., can be terminated with medical intervention, but does not terminate spontaneously) at time of enrollment
* Patient is in cardiogenic shock defined by systolic blood pressure < 90 mmHg and on pressor/inotrope medications at time of potential enrollment
* Patient has 2 or 3 degree heart block at time of potential enrollment
* Patient has undergone or is scheduled for a coronary artery bypass graft procedure, 30 days before or 30 days after date of potential enrollment
* Patient has a known life expectancy of less than 6 months due to non cardiac causes
* Patient has marked renal dysfunction defined as Creatinine > 2.5 mg/dL at time of enrollment
* Patient enrolled in any concurrent study that may confound the results of the study
* Patient is in class IV heart failure
* Patient is on the heart transplant list
* Patient already has an implanted pacemaker, ICD, or CRT device
* Patient is pregnant or plans to be pregnant during the course of the study
* Both

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2005-05 (Actual); Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
LVEDV | 12 months

SECONDARY OUTCOMES:
LVESV | 12 months
ECG | 12 months
Blood chemistry | 12 months
Device parameters | 12 months
Quality of Life | 12 months
Cardiac echo | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Chung, MD, Principal Investigator — Christ Hospital Cincinnati
Locations (1):
- Christ Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chung ES, Dan D, Solomon SD, Bank AJ, Pastore J, Iyer A, Berger RD, Franklin JO, Jones G, Machado C, Stolen CM. Effect of peri-infarct pacing early after myocardial infarction: results of the prevention of myocardial enlargement and dilatation post myocardial infarction study. Circ Heart Fail. 2010 Nov;3(6):650-8. doi: 10.1161/CIRCHEARTFAILURE.110.945881. Epub 2010 Sep 17. PMID 20852059